CLINICAL TRIAL: NCT06447298
Title: Evaluation of the Satisfaction of Parents Accompanying Children Who Have Undergone Laparoscopic Surgery
Acronym: COELIOCOM
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0129
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Parent's Satisfaction; Pediatric Surgery; Children Laparoscopic Surgery; Coelioscopy; Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Parents accompanying children: Parents accompanying children aged 0 to 17 who have undergone laparoscopic surgery in the paediatric surgery department in Brest.
  Interventions: Other: Satisfaction questionnaires

INTERVENTIONS:
Other: Satisfaction questionnaires — Use of a post-laparoscopy satisfaction questionnaire designed to be adapted to the context of laparoscopic surgery. This post-laparoscopy questionnaire was inspired by the PedsQL generic care satisfaction questionnaire, a standardised and validated questionnaire.

SUMMARY:
An increasing number of surgeries are being performed using laparoscopic techniques. This approach significantly reduces postoperative pain and speeds up recovery. Additionally, the resulting scars are smaller compared to open surgeries. This study evaluates the quality of care and communication satisfaction among parents of children undergoing laparoscopic surgery in the pediatric surgery department of Brest. The primary goal is to assess parental satisfaction with communication during the procedure. Parents of children who have undergone laparoscopic surgery will be invited to participate. Participants will complete a satisfaction questionnaire the day after surgery and participate in a follow-up phone interview 7 to 9 days post-surgery, incorporating the child's opinion if possible.

DETAILED DESCRIPTION:
Laparoscopic surgery, also known as laparoscopy and thoracoscopy, is increasingly used in pediatric surgery. This technique involves performing procedures through small incisions using miniaturized instruments and a camera, allowing precise, real-time operation. Laparoscopy offers several advantages over traditional open surgery, such as reduced surgical trauma, shorter recovery times, smaller scars, and lower risks of complications like infections and bleeding. Despite these benefits, research on patient experience with laparoscopy is limited, particularly regarding communication between patients and healthcare teams. This study aims to assess the satisfaction of parents whose children undergo laparoscopic surgery, focusing on communication and care quality. Previous studies indicate that patient satisfaction is a critical independent measure of care quality, not necessarily linked to clinical outcomes. Enhancing patient satisfaction can also reduce postoperative complications and improve recovery.

Using a custom satisfaction questionnaire based on the standardized and validated PedsQL generic care satisfaction questionnaire, this study will evaluate parental satisfaction with communication and care regarding their child's laparoscopic surgery. Parents will complete a satisfaction questionnaire the day after surgery and participate in a follow-up phone interview 7 to 9 days post-surgery, considering the child's input if possible.Using a Likert scale, each of the 20 items in the questionnaire will be evaluated with a score between 0 (not at all satisfied) and 5 (totally satisfied). Then the sum of the scores for each item will be calculated to obtain an overall score between 0 (not at all satisfied) and 100 (totally satisfied).

The primary objective of this study is to evaluate parental satisfaction with communication after their child's laparoscopic surgery by averaging the satisfaction scores from the initial post-laparoscopy questionnaire and the follow-up telephone interview (scored from 0 to 100).

For secondary objectives, responses to open-ended questions during the telephone interview will be qualitatively analyzed to gain insights into specific aspects of the parental experience with laparoscopy. The quality of care will be assessed using scores from specific items on the questionnaires related to care quality. Additionally, the study will analyze the duration of hospitalization to explore any correlation with parental satisfaction. The evolution of satisfaction over time will be assessed by comparing initial satisfaction scores with short-term satisfaction scores obtained during the follow-up interview. This comparison aims to identify any changes in satisfaction levels, particularly concerning the post-discharge period. All data will be analyzed using descriptive statistics for frequency and mean scores, with further analysis conducted using the software Prism to ensure robustness and validity of the findings.

At the end of this study, investigators hope to identify areas for improvement in surgical care and communication, aiming to enhance the postoperative quality of life for pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Accompanying parents of children from 0 to 17 years of age
* Accompanying parents of children treated by one of the following laparoscopic procedures: laparoscopy and thoracoscopy, laparoscopies requiring a mini-laparotomy for extraction of the part, and laparoscopies carried out on an outpatient basis.
* No objection from the parent accompanying the child

Exclusion Criteria:

* Parents who are minors
* Parents under legal protection (guardianship, curatorship) or deprived of liberty
* Need for intraoperative conversion.
* Insufficient knowledge of the French language to complete the post-laparoscopy satisfaction questionnaire.
* Not affiliated to the social security system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents accompanying children undergoing laparoscopic surgery in the paediatric department in Brest.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Parent satisfaction score | day of inclusion and 7 to 9 days after laparoscopic surgery
  Mean of the 2 scores on the post-laparoscopy satisfaction questionnaires at inclusion and during the telephone interview (from 0 not at all satisfied to 100 totally satisfied). Using a Likert scale, each of the 20 items in the questionnaire will be evaluated with a score between 0 (not at all satisfied) and 5 (totally satisfied). Then the sum of the scores for each item will be calculated to obtain an overall score between 0 (not at all satisfied) and 100 (totally satisfied)

SECONDARY OUTCOMES:
Parent satisfaction | 7 to 9 days after laparoscopic surgery
  Responses to open questions about laparoscopy during the telephone interview
Quality of care | day of inclusion and 7 to 9 days after laparoscopic surgery
  Independent analysis of scores on quality of care items
Parent satisfaction | day of inclusion and 7 to 9 days after laparoscopic surgery
  Comparison of initial satisfaction (paper post-laparoscopy satisfaction questionnaire at inclusion) with short-term satisfaction (telephone call post-laparoscopy satisfaction questionnaire between the 7th and 9th day after laparoscopic surgery).
Quality of care | about 2 days
  Length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brest, Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/16614882/
- See also: Related Info — https://journals.lww.com/lww-medicalcare/abstract/1999/02000/the_pedsql___measurement_model_for_the_pediatric.3.aspx
- See also: Related Info — https://journals.lww.com/lww-medicalcare/abstract/2001/08000/pedsql__4_0__reliability_and_validity_of_the.6.aspx
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/11977437/